CLINICAL TRIAL: NCT02103686
Title: A Randomized, Open-label, 3-way Crossover Clinical Trial to Compare The Pharmacokinetics of A Pregabalin Controlled Release Tablet 300mg With Immediate Release Formulation and to Assess the Effect of High Fat Diet in Healthy Male Subjects
Brief Title: Study for Comparing The Pharmacokinetics of A Pregabalin Controlled Release Tablet 300mg With Immediate Release Formulation and to Assess the Effect of High Fat Diet in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-PRSD-1201
Record Dates: First submitted 2014-03-18; First posted 2014-04-04 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Neuropathic pain; pregabalin
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin; Drugs, Investigational

ARMS (3):
- Immediate release capsule (Active Comparator): Immediate release capsule treatment under fasted condition
  Interventions: Drug: Lyrica; Dietary Supplement: fasted
- sustained release tablet (Experimental): sustained release tablet treatment under fasted condition
  Interventions: Drug: Experimental drug; Dietary Supplement: fasted
- sustained release tablet (high fat meal) (Experimental): sustained release tablet under high fat meal condition.
  Interventions: Drug: Experimental drug; Dietary Supplement: High fat meal

INTERVENTIONS:
Drug: Lyrica
  Arms: Immediate release capsule
Drug: Experimental drug — sustained release formulation of pregabalin
  Arms: sustained release tablet; sustained release tablet (high fat meal)
Dietary Supplement: High fat meal
  Arms: sustained release tablet (high fat meal)
Dietary Supplement: fasted
  Arms: Immediate release capsule; sustained release tablet

SUMMARY:
The purpose of this study is to:

1. Compare the pharmacokinetics profiles of pregabalin sustained release tablet (300mg) to immediate release capsule(150mg * 2).
2. Evaluate the effectiveness of food to pharmacokinetics profile of Pregabalin sustained release tablet.

ELIGIBILITY:
Inclusion Criteria:

* 19~44 aged healthy adult.
* someone tho has at least 50kg body weight and ideal body weight ±20%

Exclusion Criteria:

* someone has acute symptom at screening phase
* someone has any disease or symptoms which is clinically significant
* someone had been determined during healthy examination in screening period
* AST or ALT > 1.25 times than normal
* Total bilirubin > 1.5 times than normal
* someone who has a history of allergy, anaphylaxis, drug abuse or misuse.
* someone who had enrolled to other clinical trial within the last 60 days.
* someone who had donated blood within the last 60 days.
* someone who can't take a meal derived from this trial.
* someone who has taken abnormal meals like which can affect to drug ADME
* someone who has taken other ETC drugs or oriental drugs within the last 14 days, Or OTC drugs within the last 7 days
* someone who has taken caffein continuously (coffee or green tea more than 5 cups per a day) or took caffein since 24hours before.
* someone who has taken alcohol more than 30g/day or smoked more than 10 piece of tobacco/day.
* someone who has galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cmax, AUC of pregabalin | 0~36h

SECONDARY OUTCOMES:
Safety evaluation | 0~24day